CLINICAL TRIAL: NCT03313999
Title: Measuring Skin Elasticity in Lymphedema Patients
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Device was unable to be serviced
Sponsor: Beth Israel Deaconess Medical Center (Other)
Responsible Party: Principal Investigator, Dhruv Singhal, Associate Professor, Beth Israel Deaconess Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2024P000442
Record Dates: First submitted 2017-10-14; First posted 2017-10-19 (Actual); Last update posted 2025-10-20 (Actual); Status verified 2025-10

CONDITIONS: Diagnoses Disease; Lymphedema
Keywords: Lymphedema indentometer; Durometer
MeSH Terms: conditions — Lymphedema

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Durometer Measurement (Other): All patients participating in the study will receive standard of care treatment for their lymphedema. As part of the study they will be measured by the durometer in addition to other, standard diagnostics to further characterize their lymphedema progression.
  Interventions: Device: Lymphedema Indentometer

INTERVENTIONS:
Device: Lymphedema Indentometer — The subject will sit down. The machine will be placed over their extremity/affected region. They will then be told the machine will be activated. They may or may not feel the machine touch them. A small pressure will be applied to the skin surface for 4 seconds. The computer will record the skin elasticity as change in resistance to compression over time during these 4 seconds. The entire procedure will take about a minute or less, after which the standard of care visit with the physical therapist will continue.
  Other Names: Durometer

SUMMARY:
This protocol will utilize the lymphedema indentometer, or durometer (a novel, noninvasive piece of equipment that measures skin elasticity), to better characterize disease progression in patients with lymphedema. Beth Israel Deaconess Medical Center patients who undergo treatment of lymphedema will be candidates for this noninvasive test. This device and the data it generates will help understand the incidence of lymphedema at Beth Israel Deaconess Medical Center compared to national data and the outcomes of surgical treatment of lymphedema.

ELIGIBILITY:
Inclusion Criteria:

* Patients evaluated by the Beth Israel Deaconess Medical Center Lymphedema team with a diagnosis of lymphedema OR determined to be at risk of developing Lymphedema in any of their extremities
* Patients must be over 18 years of age
* Patients must be willing and capable to provide informed consent
* Patients must speak English

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2018-02-18 (Actual); Primary Completion 2025-06-02 (Actual); Study Completion 2025-06-02 (Actual)

PRIMARY OUTCOMES:
Durometer Measurement | Enrollment (3 years)
  Value providing measure for the viscoelastic properties of skin including firmness and mechanical creep.

CONTACTS AND LOCATIONS:
Overall Officials: Dhruv Singhal, MD, Principal Investigator — Beth Israel Deaconess Medical Center
Locations (1):
- Beth Israel Deaconess Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
Data from this study's data repository may be accessed by investigators interested in using the repository for research purposes. To access the data, investigator(s) will need to obtain Institutional Review Board approval of their protocol and submit their protocol to Dhruv Singhal, MD for review. Dr. Singhal will review the request for feasibility, scientific validity, and proper regulatory approvals. Only once the investigator(s) have received written Institutional Review Board approval, written approval from Dr. Singhal, and, if necessary, completed a material transfer agreement will they be given access to data from the repository. Dr. Singhal is uniquely suited to review requests to use repository data as he is a pioneer in the study and treatment of lymphedema and familiar with all information contained in the database.
Supporting Information: Study Protocol
Time Frame: Researchers will only have access to information in the study's database for the duration of their Institutional Review Board approval.
Access Criteria: After the interested investigator(s) receive Institutional Review Board approval and approval from Dr. Singhal, the study team will securely send the data to the requesting investigator. Any requesting investigator will receive only durometer measurements, lymphedema characteristics and demographic information from the database. In all cases the requesting investigator will receive only de-identified data.